CLINICAL TRIAL: NCT05689853
Title: An Open-label, Multicenter, Phase Ib/II Study to Evaluate the Safety, Tolerability and Antitumor Activity of AK119 in Combination With AK112 in Patients With Advanced Solid Tumors
Brief Title: Study of AK119 Combined With AK112 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ak119-105
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK119 in combination with AK112 (Experimental): AK119 and AK112, IV, every 3 weeks
  Interventions: Drug: AK119; Drug: AK112

INTERVENTIONS:
Drug: AK119 — AK119 is an anti-CD73 monoclonal antibody.
Drug: AK112 — AK112 is a bispecific monoclonal antibody against VEGF and PD-1.

SUMMARY:
This is a Phase Ib/II study to assess the safety, tolerability and preliminary efficacy of AK119 combined with AK112 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily written informed consent and agree to comply with all protocol-specified procedures and follow-up evaluations
2. Age ≥ 18 years and ≤ 75 years
3. Histologically or cytologically-confirmed diagnosis of advanced/unresectable solid tumor that have been progressed or intolerant to at least one standard treatment regimen in the advanced or metastatic setting, if such a therapy exists
4. Measurable lesion based on RECIST v1.1
5. ECOG status of 0 or 1
6. Life expectancy ≥ 3 months
7. Adequate organ function
8. Women of childbearing potential and men with female partners of childbearing potential must agree to use effective contraception during treatment and for at least 120 days following the last dose of study treatment

Exclusion Criteria:

1. Known other active malignancy within 3 years prior to the first dose of investigational product, with the exception of early stage cancers that have treated with curative intent
2. Currently participating in another study unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study
3. Received systemic antineoplastic therapy ( e.g. chemotherapy, radiotherapy, immunotherapy) within 4 weeks prior to the first dose of investigational product; received small-molecule anticancer agents within 2 weeks prior to the first dose of investigational product
4. In addition to anti-PD-(L)1 monoclonal antibody, prior exposure to other immune checkpoint inhibitors or any other treatment directed to tumor immune mechanism
5. Prior therapy targeting CD73 or CD39 or the adenosine signalling pathway
6. Treatment with non-steroidal anti-inflammatory drugs, anti-platelet agents or anticoagulants within 7 days prior to the first dose of investigational product
7. Current dependency on systemic therapy with glucocorticoids (>10 mg/day prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of investigational product
8. Presence of spinal cord compression or active brain metastases
9. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage
10. History or presence of a serious hemorrhage or known bleeding tendency within 3 months
11. Active autoimmune disease that has required systemic treatment in past 2 years
12. Clinically significant cardiovascular disease
13. History of interstitial lung disease or noninfectious pneumonitis
14. Received systemic anti-infective therapy (excluding antiviral therapy for hepatitis B or C) within 14 days prior to the first dose of investigational product
15. Major surgical procedure or serious trauma within 28 days prior to the first dose of investigational product
16. History of immunodeficiency, human immunodeficiency virus infection (HIV)
17. Active tuberculosis or syphilis infection
18. History of organ transplantation or allogeneic haematopoietic stem cell transplantation
19. Toxicities of prior anticancer therapy have not resolved to ≤ Grade 1 (NCI-CTCAE version 5.0)
20. Any other conditions that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | During the first three weeks
  DLTs will be assessed during the first three weeks of treatment. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug.
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with CR or PR (based on RECIST Version 1.1).

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1).
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST Version 1.1).
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to 2 years
  Time to response (TTR) is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR (based on RECIST Version 1.1).
Time to progression (TTP) | Up to 2 years
  Time to progression (TTP) is defined as the time from the start of the treatment to the documentation of disease progression (based on RECIST Version 1.1).
Overall survival (OS) | Up to 2 years
  OS defined as the time from the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Wu, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China